CLINICAL TRIAL: NCT06492512
Title: Oral Iron Supplementation on Alternate Vs. Consecutive Days for Iron Deficiency Anemia in Pregnancy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-924
Record Dates: First submitted 2024-06-28; First posted 2024-07-09 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-07

CONDITIONS: Iron-deficiency Anemia (IDA); Pregnancy
Keywords: Iron-deficiency anemia (IDA); Iron-deficiency anemia (IDA) during gestation
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 for daily iron (ferrous sulfate) supplementation vs. every other day iron (ferrous sulfate) supplementation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1) Daily dose of ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill (Experimental): daily (Group 1) supplementation with one oral pill containing ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill
  Interventions: Drug: daily ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill
- 2) Alternate daily dose of ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill (Experimental): alternate day (Group 2) supplementation with one oral pill containing ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill
  Interventions: Drug: alternate day ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill

INTERVENTIONS:
Drug: daily ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill — ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill daily
  Other Names: daily
  Arms: 1) Daily dose of ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill
Drug: alternate day ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill — ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill every other day
  Other Names: alternate day
  Arms: 2) Alternate daily dose of ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill

SUMMARY:
This will be a randomized clinical trial. Enrolled subjects will be randomized (1:1) into two study arms to receive either daily (Group 1) or alternate day (Group 2) supplementation with one oral pill containing ferrous sulfate with an equivalent elemental iron dose of 65 mg per pill.

DETAILED DESCRIPTION:
During the enrollment (baseline) visit, subjects will undergo a blood draw to assess hemoglobin, ferritin and soluble transferrin receptor (sTfR) levels to confirm current depleted iron stores and will then be randomly allocated into one of the two study arms. All ferrous sulfate (oral tablets) will be provided to patients by the investigators. All subjects will be instructed to take oral iron on an empty stomach or 1 hour after meals for better absorption, preferably with a vitamin C rich product such as orange juice. To minimize variability introduced by other potential iron sources, prenatal vitamins that have the same amount and form of iron will be provided to both study groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients will be enrolled at less than 30 weeks gestational age (GA) with laboratory confirmed IDA (as defined by hemoglobin under 10.5 g/dL, as well as ferritin under 15 mcg/L)

Exclusion Criteria:

* Patients <18 years old, patients who have severe IDA that requires blood transfusion or IV iron infusion, patients who have other known hemoglobinopathy (such as thalassemia or sickle cell anemia) or anemia of different mechanism (such as vitamin B12 or folate deficiency), patients with ulcerative colitis, Crohn's disease, gastric ulcers, patients who have previously undergone gastric bypass surgery, patients who experience admission for antepartum bleed, have been diagnosed with abnormal placentation (i.e., placenta previa, placenta accreta, placenta increta or percreta)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 120 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
reversal of iron deficient anemia | 8 weeks after the baseline visit ± 7 days
  hemoglobin > 10.5 g/dL
reversal of iron deficient anemia | 8 weeks after the baseline visit ± 7 days
  ferritin > 15 mcg/L

SECONDARY OUTCOMES:
soluble transferrin receptor (sTfR) levels within normal range | 8 weeks after the baseline visit ± 7 days
  1.8-4.6 mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Yahia Zeino, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No